CLINICAL TRIAL: NCT01184937
Title: Effect of Patient Education on Kidney Recipients Knowledge, Coping and Quality of Life. A Randomized Controlled Trial.
Brief Title: Effect of Patient Education on Kidney Recipients Knowledge, Coping and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 182014/V52
Record Dates: First submitted 2010-06-25; First posted 2010-08-19 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Renal Recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient education program (Experimental)
  Interventions: Behavioral: Patient education program
- Standard care (No Intervention)

INTERVENTIONS:
Behavioral: Patient education program — All patients receive standard care. Experimental group receive a structured patient education program based in self-care theory and pedagogical theory, build upon the the principles of the "Pro-Self education program". The intervention program consist of five weekly one-to-one sessions with a transplant nurse, lasting about 40-60 minutes, starting during the first week after discharge and lasting until 7 weeks post transplantation. Education content consists of two levels: general knowledge level and individual knowledge. Each session has a specific program. In addition, academic detailing is used to describe patient's knowledge levels and for tailoring the education to individual needs.
  Arms: Patient education program

SUMMARY:
For patients with end-stage kidney disease, transplantation is the treatment of choice, offering improved quality of life by restored metabolism and freedom from dialysis. However, demands regarding the acquirement of knowledge in life post transplantation are high. In order to reduce rejection episodes, graft loss and the negative consequences of life-long immunosuppressive medication, it is essential for kidney recipients to possess knowledge about important aspects regarding immunosuppressive medication, graft surveillance and the benefit of specific lifestyle behavior. Consequently, patient education is required for this patient group. This randomized controlled trial is investigating the effect of a structured patient education program on kidney recipients' knowledge, coping and quality of life

ELIGIBILITY:
Inclusion Criteria:

* being over 18
* recently had a kidney transplant
* able to speak, understand and read Norwegian
* mentally able to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Kidney recipients'knowledge level | 7-8 weeks post kidney transplantation
  Knowledge level is measured by a self-administrated knowledge questionnaire consisting of 19 items addressing knowledge in relation to three areas: medication, rejection and lifestyle. Each item is rated using a 5 points scale, anchored on the left with the wording "totally disagree"(1), "rather disagree" (2) "either agree or disagree" (3), "quite agree" (4) and to the left with "totally agree"(5). Patients are asked to put a ring around a number to indicate their level of agreement with each item.
Kidney recipients'knowledge level | 6 months post kidney transplantation
  Knowledge level is measured by a self-administrated knowledge questionnaire consisting of 19 items addressing knowledge in relation to three areas: medication, rejection and lifestyle. Each item is rated using a 5 points scale, anchored on the left with the wording "totally disagree"(1), "rather disagree" (2) "either agree or disagree" (3), "quite agree" (4) and to the left with "totally agree"(5). Patients are asked to put a ring around a number to indicate their level of agreement with each item.

SECONDARY OUTCOMES:
Kidney recipients' coping | 7-8 weeks post kidney transplantation
  Coping is measured by the following self-administrated questionnaires: "The Generalized Self-efficacy Scale", "The Long-term Medication Behavior Self-efficacy Scale" and "The Moriscy Compliance scale". In addition, the number of missing observations in the patients' "transplant diaries" is counted.(The "transplant diary" contains patients own daily observations of graft function and signs of rejection). Number of missing observations are counted from observation start and during a period of 7-8 weeks. The percent of missed observations of total possible observations are estimated.
Kidney recipients' coping | 6 months post kidney transplantation
  Coping is measured by the following self-administrated questionnaires: "The Generalized Self-efficacy Scale", "The Long-term Medication Behavior Self-efficacy Scale" and "The Moriscy Compliance scale".
Kidney recipients' quality of life | 7-8 weeks post kidney transplantation
  Quality of life is measured by the following self -adminstred questionnaires: The acute version of the "Short Form Health Survey" (SF-12) and the disease-spesific quality of life questionnaire: "The Kidney Transplant Questionnaire"
Kidney recipients' quality of life | 6 months post kidney transplantation
  Quality of life is measured by the following self -adminstred questionnaires: The acute version of the "Short Form Health Survey" (SF-12) and the disease-spesific quality of life questionnaire: "The Kidney Transplant Questionnaire"

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829